CLINICAL TRIAL: NCT04745312
Title: The Effect of Lighting Supplementation on Cognitive Task Performance During the Day
Brief Title: Effect of Lighting Supplementation on Daytime Cognition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shadab A Rahman, Associate Neuroscientist, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2019P000900; 2020A011565 (Other Grant/Funding Number: Biological Innovation and Optimization Systems, LLC.)
Record Dates: First submitted 2021-02-04; First posted 2021-02-09 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Non-visual Effects of Light
Keywords: Light; Cognition; Alertness; Learning

STUDY DESIGN:
Intervention Model Description: Randomized crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ambient light (Active Comparator): Fluorescent ambient lighting
  Interventions: Device: Visible light
- Ambient light plus task lamp (Experimental): Fluorescent ambient lighting plus task lamp
  Interventions: Device: Visible light

INTERVENTIONS:
Device: Visible light — Ambient room lighting will be supplemented with additional light from a task lamp.

SUMMARY:
The aim of the study is to examine the efficacy of supplementing sub-optimal ambient room lighting with a task lamp on working memory and procedural learning.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-30 years;
* Healthy (no medical, psychiatric or sleep disorders;
* Non-smoking for at least 6 months;
* Body Mass Index of >18 or <30 kg/m2;
* Able to maintain 7-hour consistent sleep schedule during the study
* Able to refrain from caffeine, alcohol, medication and supplements during the study

Exclusion Criteria:

* History of alcohol or substance abuse;
* positive result on drugs of abuse urine toxicology;
* Current or past history of sleep disorders, including but not limited to obstructive sleep apnea, narcolepsy, insomnia, or any significant sleep complaint
* Psychiatric disorder, or first degree relative with a psychiatric disorder
* Recent acute or chronic medical disorder
* Use of drugs or medication (birth control OK) likely to affect sleep, alertness or light sensitivity, as determined by the investigators
* Visual disorder, including but not limited to color blindness, or family history of glaucoma
* Pregnancy or lactation
* Shift work (> 2 nights / week in the last 3 months and not during the study)
* Transmeridian travel (2 or more time zones) in the past 3 months
* Any other reason as determine by the Principal Investigator

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Working memory | 8 hour light exposure
  Percent correct responses on a 2-minute mental arithmetic task

SECONDARY OUTCOMES:
Procedural learning | 8 hour light exposure
  Percent change in the number of correct sequences on the Motor Sequence Task

OTHER OUTCOMES:
Vigilance | 8 hour light exposure
  Reaction time and lapses on the Psychomotor Vigilance Task
Subjective sleepiness | 8 hour light exposure
  Subjective sleepiness assessed by the Karolinska Sleepiness Scale - Scale from 1-9 where higher scores indicate greater sleepiness
Memory recall | 8 hour light exposure
  Percentage of correctly recalled words on a paired associates task
Psychological distress | 8 hour light exposure
  Total score on the Profile of Mood States (POMS)
Affect | 8 hour light exposure
  Positive and negative affect scores assessed by the PANAS

CONTACTS AND LOCATIONS:
Overall Officials: Shadab A Rahman, PhD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grant LK, Crosthwaite PC, Mayer MD, Wang W, Stickgold R, St Hilaire MA, Lockley SW, Rahman SA. Supplementation of ambient lighting with a task lamp improves daytime alertness and cognitive performance in sleep-restricted individuals. Sleep. 2023 Aug 14;46(8):zsad096. doi: 10.1093/sleep/zsad096. PMID 37026184